CLINICAL TRIAL: NCT02727270
Title: Measuring Cortisol Levels in Persons With Parkinson's (PD)
Acronym: CORT-PD
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency); Oregon Clinical and Translational Research Institute (Other); Huntington's Disease Society of America (Other)
Responsible Party: Principal Investigator, Amie Hiller, MD, Neurologist, Oregon Health and Science University
Other Study IDs: 15183; 3794 (Other: VA Portland Health Care System); 5338 (Other: Oregon Clinical Translational Research Institute); 4546 (Other: VA Portland Health Care System); 7186 (Other: Oregon Clinical Translational Research Institute)
Record Dates: First submitted 2016-03-21; First posted 2016-04-04 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease; Huntington Disease
Keywords: Movement disorders; Metabolic Stress; Basal Ganglia Disorders
MeSH Terms: conditions — Parkinson Disease; Huntington Disease; Movement Disorders; Basal Ganglia Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Parkinson's - High Stress *FULL NOT RECRUITING: Parkinson's disease patients with self-reported high strain/stress.
  Interventions: Other: No Intervention - Observational Study
- Parkinson's - Low Stress *FULL NOT RECRUITING: Parkinson's disease patients with self-reported low strain/stress.
  Interventions: Other: No Intervention - Observational Study
- Controls - High Stress *FULL NOT RECRUITING: Healthy controls (no neurological disease) with self-reported high strain/stress.
  Interventions: Other: No Intervention - Observational Study
- Controls - Low Stress *FULL NOT RECRUITING: Healthy controls (no neurological disease) with self-reported low strain/stress.
  Interventions: Other: No Intervention - Observational Study
- Huntington's - High Stress *FULL NOT RECRUITING: Huntington's disease patients and/or Huntington's disease gene carriers with self-reported high strain/stress.
  Interventions: Other: No Intervention - Observational Study
- Huntington's - Low Stress *FULL NOT RECRUITING: Huntington's disease patients and/or Huntington's disease gene carriers with self-reported low strain/stress.
  Interventions: Other: No Intervention - Observational Study
- Parkinson's Disease - ReEnrollment (COVID-19) *FULL NOT RECRUITING: Parkinson's disease patients that had previously completed the study.
  Interventions: Other: No Intervention - Observational Study

INTERVENTIONS:
Other: No Intervention - Observational Study — No Intervention - Observational Study

SUMMARY:
The objective of this study is to evaluate the cortisol awakening response with persons with Parkinsons Disease (PD), Huntingtons Disease (HD), and controls. These data are desired so experience can be gained with measuring stress levels subjectively and objectively in persons with PD, HD, and controls.

DETAILED DESCRIPTION:
Telephone consent will be obtained.

Participants will collect saliva at twelve time points - four times a day for three days.

Visits will be conducted virtually (over the internet).

The virtual visit is to assess Parkinson's or Huntington's disease status, stress, mood, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Group (3) Inclusion:

* No significant neurological disorder
* PSS score of greater than or equal to 13.

Group (5) Inclusion:

* HD diagnosis or HD gene carrier
* a Perceived Stress Scale (PSS) score higher than or equal to 13.

Group (6) Inclusion:

* HD diagnosis or HD gene carrier
* PSS score lower than 13

Group (7) Inclusion:

* PD diagnosis
* Prior completion of the study.

Exclusion Criteria:

* The use of medications known to effect cortisol levels (estrogen, synthetic glucocorticoids, androgens, phenytoin, spironolactone, prednisone, prednisolone, and hydrocortisone).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll seven groups: (1) person with PD and moderate levels of self-reported stress, (2) persons with PD and low levels of self-reported stress, (3) controls and moderate levels of self-reported stress, (4) controls and low levels of self-reported stress, (5) persons with HD and moderate/high levels of self-reported stress, and (6) persons with HD a low levels of self-reported stress, and (7) those that completed the study prior to COVID-19 restrictions in March of 2020.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-06; Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Awakening Salivary Cortisol level (ug/dL) Response | Collected upon awakening and 30 minutes after awakening
  Salivary Cortisol level (ug/dL) Response is the change in cortisol between awakening and 30 minutes after awakening.

CONTACTS AND LOCATIONS:
Overall Officials: Amie L Hiller, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science Universtiy, Portland, Oregon
  - VA Portland Health Care System, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data be available (including data dictionaries). Individual participant data that underlie the results reported the resultant article, after deidentification (text, tables, figures, and appendices). In addition to data, the study protocol and the informed consent form (ICF) will be provided. Data will be available beginning 6 months and ending 2 years following article publication.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months - 2 years following article publication
Access Criteria: Data will be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Data will be released to achieve aims in the approved proposal or for individual participant data meta-analysis.
URL: https://www.parkinsons.va.gov/northwest/

REFERENCES:
- [Background] Ceravolo R, Frosini D, Poletti M, Kiferle L, Pagni C, Mazzucchi S, Volterrani D, Bonuccelli U. Mild affective symptoms in de novo Parkinson's disease patients: relationship with dopaminergic dysfunction. Eur J Neurol. 2013 Mar;20(3):480-485. doi: 10.1111/j.1468-1331.2012.03878.x. Epub 2012 Oct 18. PMID 23078376
- [Background] Hartmann A, Veldhuis JD, Deuschle M, Standhardt H, Heuser I. Twenty-four hour cortisol release profiles in patients with Alzheimer's and Parkinson's disease compared to normal controls: ultradian secretory pulsatility and diurnal variation. Neurobiol Aging. 1997 May-Jun;18(3):285-9. doi: 10.1016/s0197-4580(97)80309-0. PMID 9263193
- [Background] Marsden CD, Owen DA. Mechanisms underlying emotional variation in parkinsonian tremor. Neurology. 1967 Jul;17(7):711-5. doi: 10.1212/wnl.17.7.711. No abstract available. PMID 6067490
- [Background] Matousek RH, Dobkin PL, Pruessner J. Cortisol as a marker for improvement in mindfulness-based stress reduction. Complement Ther Clin Pract. 2010 Feb;16(1):13-9. doi: 10.1016/j.ctcp.2009.06.004. Epub 2009 Jul 4. PMID 20129404